CLINICAL TRIAL: NCT06678867
Title: A Phase II Multicentre Trial for the Use of 5-ALA Paediatric Patients With High Grade Brain Tumours
Brief Title: The Use of 5-ALA in Paediatric Patients With High Grade Brain Tumours
Acronym: P5A
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UCL/154416; CCLGA 2022 27 Dandapani (Other Grant/Funding Number: Little Princess Trust- Children's Cancer and Leukaemia Group)
Record Dates: First submitted 2024-10-28; First posted 2024-11-07 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Brain Tumor
Keywords: Ependymoma; Glioma; Paediatric; 5-ALA; Brain tumour
MeSH Terms: conditions — Brain Neoplasms; Ependymoma; Glioma

STUDY DESIGN:
Intervention Model Description: This is a phase II, multicentre, non-randomised open-label trial with two cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with high grade brain tumours (Other): This is a single-arm study with two cohorts
  Interventions: Drug: 5-ALA (Gliolan)

INTERVENTIONS:
Drug: 5-ALA (Gliolan) — Gliolan 30 ml/mg powder for oral solution, Single dose 3-6 hours prior to surgery

SUMMARY:
The aim of the study is to examine the safety and feasibility of using 5-ALA in children who have MRI scans showing an aggressive looking brain tumour. It will also study if 5-ALA can help the surgeon achieve maximal tumour removal and discriminate between normal brain tissue and tumour.

Patients will be between 3-18 years (inclusive) and all patients will receive 5-ALA 3-6 hours prior to resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Magnetic Resonance Imaging confirmation of diagnosis consistent with either: primary presentation of high grade brain tumour OR patient relapsing with previously confirmed ependymoma or high-grade glial tumour
* Tumours will be either intrinsic supratentorial or infratentorial / posterior fossa, non-brainstem, tumours
* Patient is appropriate for maximal safe resection of tumour, based on Investigator and Multidisciplinary Team judgement
* 3 - 18 years inclusive
* Adequate liver and kidney function

  * creatinine - less than one and a half times the upper limit of normal.
  * haemoglobin above the lower limit of normal
  * Alanine transferase or Aspartate transferase less than twice the upper limit of normal (if both performed, then both results must be lower than twice the upper limit of normal
  * bilirubin lower than one and a half times the upper limit of normal
* Normal Coagulation profile

  o Prothombin Time, Activated Partial Prothombin Time and Thrombin Time all within normal limits
* Urine porphyrin - Test to be completed and sent for analysis
* Blood pressure lower than or equal to the upper limit of normal
* Negative pregnancy test in women of childbearing potential*
* Informed Consent *A positive pregnancy test that is suspected to be due to the location of the tumour is to be queried with the TMG prior to registration of the patient

Exclusion Criteria:

* Patients with low grade tumours (either radiological or histological diagnosis)
* Patient is appropriate for biopsy only, based on Investigator and MDT judgement
* Known history (including family history) of porphyria
* Hypersensitivity to the active substance or to porphyrins
* History of light sensitivity reactions
* Pregnant or breastfeeding women

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Complete resection rate and fluorescence rate of supratentorial instrinsic high grade brain tumours. Cohort 2: Fluorescence rate of infratentorial tumours. | Two weeks
  Timeframe between informed consent and surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Children's Hospital, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Following data protection guidance